CLINICAL TRIAL: NCT04211168
Title: Toripalimab Plus Lenvatinib as Second-line Treatment in Advanced Biliary Tract Cancers: a Single-arm, Non-randomized, Single-center Clinical Trial and Biomarker Study
Brief Title: Toripalimab Plus Lenvatinib as Second-line Treatment in Advanced Biliary Tract Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-2171
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-10

CONDITIONS: Advanced Biliary Tract Cancer
Keywords: Intrahepatic cholangiocarcinoma; hilar cholangiocarcinoma; common bile duct cancer; gallbladder cancer; Toripalimab; Lenvatinib; biomarker
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor; Gallbladder Neoplasms | interventions — toripalimab; lenvatinib

STUDY DESIGN:
Intervention Model Description: Patients are confirmed with advanced biliary tract cancers by imaging and histological examination and meet with the inclusive criteria, including intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, common bile duct cancer and gallbladder cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Plus Lenvatinib (Experimental): Toripalimab (Shanghai Junshi Biosciences Co., Ltd.) is a recombinant anti-human PD-1 IgG4 monoclonal antibody.
  Lenvatinib is a novel angiogenesis inhibitor which targets multiple tyrosine kinases， including vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β, RET and KIT.
  Interventions: Drug: Toripalimab plus Lenvatinib

INTERVENTIONS:
Drug: Toripalimab plus Lenvatinib — Toripalimab 240mg, every 3 weeks, intravenous infused, day 1, 6 weeks a cycle.
  Lenvatinib 8mg (weight<60kg) or 12mg (weight≥60kg), once a day, orally, day 2, 6 weeks a cycle. Dose reduction to 4mg/d or dose termination is allowed according to adverse events.
  Number of cycle: until progression or unacceptable toxicity events develop.
  Other Names: JS001 plus E7080

SUMMARY:
The investigators design a phase II clinical study to explore the efficacy and safety of toripalimab plus lenvatinib as a second-line treatment in patients with advanced biliary tract cancers and to analyze potential biomarkers of therapeutic response.

DETAILED DESCRIPTION:
This phase II trial is a single-arm, non-randomized and single-center clinical study.

It is estimated that 44 patients who met the study criteria will be enrolled in 2 years and treated with toripalimab plus lenvatinib in PUMCH. The investigators will follow up and collect subjects' data each month to evaluate the efficacy and safety of treatment, including overall survival and time to progression, until disease progression or death. Interim analysis and final analysis will be conducted when collecting data from 20 and 44 subjects, respectively in this trial. Histopathology and multi-omics data analysis will be used to explore potential biomarkers of treatment response.

Study Type: Interventional.

Masking: Open Label.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following criteria

* Subjects volunteer to participate in the study and agree to sign the informed consent with good compliance and follow-up.
* Subjects are 18 years old or older when signing the informed consent and gender is not limited.
* Subjects were diagnosed with advanced biliary tract cancers by imaging and histological examination, including intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, common bile duct cancer and gallbladder cancer. Advanced biliary tract cancers refer to unresectable, recurrent, locally advanced and metastatic lesions which are defined as stage IIIA or above according to the 8th AJCC stage system.
* The disease is not suitable for radical surgery and/or topical treatment, or disease progression occurs after surgery and/or local treatment, including lesion resection, ablation, transcatheter arterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC), radiotherapy at least 4 weeks before the baseline assessment. All acute toxic effects of local treatment must be ≤ CTCAE 5.0 Level 1.
* Patients are intolerant or fail after first-line systemic treatment (gemcitabine or platinum based regimen) and require palliative treatment. The first-line system treatment failure was ≥ 1 month before enrollment in this study (signing informed consent) and adverse events are controlled (NCI-CTCAE ≤ Grade Ⅰ). i) Definition of systemic treatment: Gemcitabine or platinum based regimen for more than 1 cycle. Adjuvant chemotherapy based on gemcitabine or platinum is considered as first-line treatment if recurrence occur during or after 6 months adjuvant chemotherapy sequential to tumor resection. ii) Definition of treatment failure: Disease progression occur during treatment or in 6 months after the last cycle. iii) Definition of intolerance: Grade ≥IV hematologic toxicity; grade ≥III toxicity of liver, kidney and skin; grade ≥ II toxicity of heart, lung and brain.
* Prior treatment must not include lenvatinib, PD-1 / PD-L1 antibodies or molecular targeted therapy for ≥ 14 days.
* At least one measurable lesion (according to RECIST version 1.1): the measurable lesion has a long diameter ≥ 10 mm or lymphadenopathy has a short diameter ≥ 15 mm in spiral CT scan.
* Blood pressure is controlled <= 150/90 mmHg with no more than 3 antihypertensive drugs.
* The ECOG score is 0-1 within 1 week before enrollment.
* Estimated survival time ≥ 12 weeks.
* Liver function assessment: Child-Pugh Grade A or mild Grade B (score ≤ 7).Only one of albumin and bilirubin is Child-Pugh score 2.
* Patients with active hepatitis B and C need to receive relevant antiviral treatment. HBV DNA <2000 IU/ml (10^4 copies/ml) and HCV-RNA negative.
* No more than 2 organs metastasis, including liver, lung, bone and brain.
* Hematology and organ function are well based on the following laboratory results within 14 days prior to the treatment of this study: i) Whole blood cell examination (no blood transfusion within 14 days, no G-CSF use and no drugs use): Hb≥100g/L, ANC≥1.5×10*9/L, PLT≥75×10*9/L. ii) Biochemical examination (no ALB infused within 14 days): ALB≥30g/L, ALT, AST and ALP<5×ULN, TBIL≤60 μmol/L, creatinine≤1.5×ULN or CCr >50mL/min. iii) Coagulation function: International standardized ratio (INR) ≤ 1.5 × upper limit of normal (ULN), or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; or PT ≤ULN + 4s.
* No active autoimmune diseases that require systemic therapy in the past 2 years (note: active state means requiring disease modulators, corticosteroids or immunosuppressive drugs use). Alternative therapies, such as thyroxine, insulin or a physiological corticosteroid replacement therapy are not considered as systemic therapy.
* Women with fertility agree to abstinence during the treatment period and at least 6 months after the last dose (avoiding heterosexual intercourse) or using a contraceptive method with an annual contraceptive failure rate <1%. i)If a female patient has menstruation and not reached the postmenopausal state (continuously no menstruation ≥ 12 months and no other causes), and has not undergone sterilization by removing the ovaries and/or uterus), then the patient has fertility. ii) Contraceptive methods with a contraceptive failure rate <1% include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices. iii) The reliability of sexual desire should be evaluated relative to the duration of the clinical trial and lifestyle of patient. Periodic abstinence (eg. calendar days, ovulation, symptomatic body temperature or post-ovulation methods) and in vitro ejaculation are unacceptable methods of contraception.
* Male patients agree to abstinence (no heterosexual intercourse) or use of contraceptive measures and no sperm donation, as defined below: i) When a female partner has fertility, male patients must abstinence from sex during treatment and at least 6 months after the last dose of treatment, or use condoms and other contraceptive methods with contraceptive failure rate <1%. At the same time, male patients must also agree not to donate sperm. ii) When a female partner is pregnant, the male patient must abstinence or using a condom during the treatment period and at least 6 months after the last dose of treatment to prevent the fetus from being affected by the study. iii) The reliability of sexual desire should be evaluated relative to the duration of the clinical trial and lifestyle of patient. Periodic abstinence (eg. calendar days, ovulation, symptomatic body temperature or post-ovulation methods) and in vitro ejaculation are unacceptable methods of contraception.
* Tumor tissue must be available for biomarker analysis prior to the first dose of treatment, If not available, participants can consult the investigator for enrollment agreement.

Exclusion Criteria: Subjects with one or more than one of the following criteria should be excluded

* Patients meet with any of the following condition: Suitable for radical surgery; Or, without an assessment lesion after radical surgery; Or, never receive any first line treatment.
* Patients who received first-line chemotherapy within 1 month when participating in the study.
* Already known to be allergic or intolerant to recombinant humanized PD-1 monoclonal antibody drugs (or components) or lenvatinib.
* Previously received with lenvatinib, or any anti-vascular endothelial growth factor (VEGF) or VEGF receptor targeted drug, or any anti-PD-1, anti-PD-L1 or anti-PD-L2 or CTLA-4 drug, including antibodies involved in JS001 clinical studies.
* ECOG score ≥ 2 points.
* Hepatic encephalopathy.
* Histopathological result show mixed liver cancer, squamous cell carcinoma or sarcoma cell component.
* More than 2 organs metastasis, including liver, lung, bone and brain.
* pregnant women (positive pregnancy test before taking the drug) or lactating women.
* Patients with bone metastases who had received palliative radiotherapy within 4 weeks before participating in the study (radiotherapy area>5% bone marrow area).
* Received any topical treatment within 4 weeks prior to the study, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection.
* Received any systemic anti-tumor treatment within 3 months prior to participation in the study, including but not limited to intravenous infused and/or oral chemotherapy, targeted drugs, antibody drugs, and traditional Chinese medicines known to have anticancer effects.
* Patients are receiving approved or developing systemic anti-cancer therapies, including chemotherapy, bio-immunotherapy, targeted therapy, or traditional Chinese medicine therapy with clear indications. Treatment received 4 weeks before randomization is permitted.
* Tumors or liver metastasis occupied more than 50% of liver volume.
* Portal vein trunk (Vp4) or inferior cavity or atrium is affected by tumor thrombus.
* Previous or existing grade 3 and above gastrointestinal fistula or non-gastrointestinal fistula (such as skin).
* Factors affect lenvatinib use, such as inability to swallow, chronic diarrhea, intestinal obstruction, or other conditions that significantly affect drug intake and absorption.
* Any >1 grade (CTC-AE5.0) unresolved toxicity due to previous treatment or operation, except for hair loss, anemia, and hypothyroidism.
* Ascites with clinical symptoms which requires abdominal puncture or drainage therapy, or Child-Pugh score >2 points.
* Hemoptysis within 4 weeks before the first medication.
* Surgery was performed within 4 weeks prior to the trial and patients must be evaluated after wound healing. Or minor surgery within 7 days before the first medication, such as simple resection and biopsy.
* Severe cardiovascular and cerebrovascular diseases, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, cerebrovascular accident or transient ischemic attack, congestive heart failure and arrhythmias within 6 months before enrollment.
* Thromboembolism (including stroke and / or transient ischemic attack) within 12 months.
* Hypertension that cannot be controlled well with antihypertensive drugs (systolic blood pressure> 150mmHg, diastolic blood pressure> 100mmHg).
* Active autoimmune disease or autoimmune disease within two years that may affect vital organ function or have/may require systemic immunosuppressive therapy. Type I diabetes, hypothyroidism requiring only hormone replacement, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss) are allowed.
* Subjects who need systemic treatment with corticosteroids (>10 mg / day prednisone or its equivalent) or other immunosuppressive drugs within 30 days of study administration. In the absence of active autoimmune disease, inhaled or topical steroids are allowed.
* Already known active central nervous system metastasis and/or cancerous meningitis. Subjects with stable brain metastases after previous treatment may participate as long as no radiologic evidence of progression lasts for at least four weeks prior to this trial and any neurological symptoms have returned to baseline, and no new or enlarged metastatic evidence in brain and no steroids use for at least 7 days prior to trial treatment. Cancer meningitis should be excluded regardless of clinical stability.
* Liver function and renal dysfunction evidence: jaundice, ascites, and/or bilirubin ≥ 60 μmol/L, proteinuria (> 3.5g /24 hours), or renal failure requiring blood dialysis or peritoneal dialysis.
* Persistent >2 grade (CTC-AE5.0) infection.
* Vaccination of any live virus vaccine within 4 weeks prior to this study.
* Biliary obstruction after clinical intervention is not remissed or needs anti-infective treatment 14 days before the first medication.
* History of allogeneic tissue transplantation or solid organ transplantation.
* History of active tuberculosis, such as mycobacterium tuberculosis.
* Female patients who are pregnant, breastfeeding or refuse contraception.
* Gastrointestinal bleeding history in the past 6 months or tendency to gastrointestinal bleeding, such as esophageal varices, local active ulceration lesions, fecal occult blood ≥ (++) (gastroscopy is required when fecal occult blood is (+)).

Evidence or history of ≥3 grade (CTC-AE5.0) bleeding events.

* History of human immunodeficiency virus infection.
* History of hepatitis B virus or hepatitis C virus infection, and not receive regular treatment.
* Severe non-healing wounds, ulcers or fractures.
* With other malignant tumors within 5 years.
* Previous and current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia and severe impairment of lung function.
* Received a potent CYP3A4 inhibitor treatment within 7 days prior to the study, or received a potent CYP3A4 inducer within 12 days prior to the study.
* There exists drug abuse, or any medical, psychological or social condition which might affect the study, the compliance or even the safety of patients.
* Informed consent can not be signed for mental or medical instability.
* Patients participate in another clinical study at the same time.
* Patients are unsuitable for participation in this research after comprehensive assessment by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | two years
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Rate of adverse events (AE) | two years
  the incidence rate of any adverse events related with treatment drugs and details include adverse events type, frequency and severity.

SECONDARY OUTCOMES:
Overall Survival (OS) | two years
  Duration from the date of initial treatment to the date of death due to any cause.
Progression-free Survival (PFS) | six months
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1) or death of any cause.
Stable Disease (SD) | two years
  Proportion of patients with stable disease status more than 4 months.
Clinical benefit rate (CBR) | two years
  Proportion of patients achieved complete response and partial response for more than 6 months.
Progression free survival rate | 6 months
  Portion of patients who do not experience disease progression (defined by RECIST 1.1) or death of any cause after treated with toripalimab plus lenvatinib for 3 months and 6 months, respectively.
6-months and 1-year mortality rate | one year
  Portion of patients who die of any cause after treated with toripalimab plus lenvatinib at 6 months and 1 year, respectively.

OTHER OUTCOMES:
Biomarkers | two years
  Any biomarker related with efficacy and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhao, MD, Study Chair — Peking Union Medical College Hospital (PUMCH)
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Banales JM, Cardinale V, Carpino G, Marzioni M, Andersen JB, Invernizzi P, Lind GE, Folseraas T, Forbes SJ, Fouassier L, Geier A, Calvisi DF, Mertens JC, Trauner M, Benedetti A, Maroni L, Vaquero J, Macias RI, Raggi C, Perugorria MJ, Gaudio E, Boberg KM, Marin JJ, Alvaro D. Expert consensus document: Cholangiocarcinoma: current knowledge and future perspectives consensus statement from the European Network for the Study of Cholangiocarcinoma (ENS-CCA). Nat Rev Gastroenterol Hepatol. 2016 May;13(5):261-80. doi: 10.1038/nrgastro.2016.51. Epub 2016 Apr 20. PMID 27095655
- [Result] Rawla P, Sunkara T, Thandra KC, Barsouk A. Epidemiology of gallbladder cancer. Clin Exp Hepatol. 2019 May;5(2):93-102. doi: 10.5114/ceh.2019.85166. Epub 2019 May 23. PMID 31501784
- [Result] Valle JW, Lamarca A, Goyal L, Barriuso J, Zhu AX. New Horizons for Precision Medicine in Biliary Tract Cancers. Cancer Discov. 2017 Sep;7(9):943-962. doi: 10.1158/2159-8290.CD-17-0245. Epub 2017 Aug 17. PMID 28818953
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Result] Valle JW, Wasan H, Lopes A, Backen AC, Palmer DH, Morris K, Duggan M, Cunningham D, Anthoney DA, Corrie P, Madhusudan S, Maraveyas A, Ross PJ, Waters JS, Steward WP, Rees C, Beare S, Dive C, Bridgewater JA. Cediranib or placebo in combination with cisplatin and gemcitabine chemotherapy for patients with advanced biliary tract cancer (ABC-03): a randomised phase 2 trial. Lancet Oncol. 2015 Aug;16(8):967-78. doi: 10.1016/S1470-2045(15)00139-4. Epub 2015 Jul 12. PMID 26179201
- [Result] Malka D, Cervera P, Foulon S, Trarbach T, de la Fouchardiere C, Boucher E, Fartoux L, Faivre S, Blanc JF, Viret F, Assenat E, Seufferlein T, Herrmann T, Grenier J, Hammel P, Dollinger M, Andre T, Hahn P, Heinemann V, Rousseau V, Ducreux M, Pignon JP, Wendum D, Rosmorduc O, Greten TF; BINGO investigators. Gemcitabine and oxaliplatin with or without cetuximab in advanced biliary-tract cancer (BINGO): a randomised, open-label, non-comparative phase 2 trial. Lancet Oncol. 2014 Jul;15(8):819-28. doi: 10.1016/S1470-2045(14)70212-8. Epub 2014 May 19. PMID 24852116
- [Result] Lamarca A, Hubner RA, David Ryder W, Valle JW. Second-line chemotherapy in advanced biliary cancer: a systematic review. Ann Oncol. 2014 Dec;25(12):2328-2338. doi: 10.1093/annonc/mdu162. Epub 2014 Apr 25. PMID 24769639
- [Result] Lamarca A, Palmer DH, Wasan HS et al. ABC-06 | A randomised phase III, multi-centre, open-label study of active symptom control (ASC) alone or ASC with oxaliplatin / 5-FU chemotherapy (ASC+mFOLFOX) for patients (pts) with locally advanced / metastatic biliary tract cancers (ABC) previously-treated with cisplatin/gemcitabine (CisGem) chemotherapy. Journal of Clinical Oncology 2019; 37: 4003-4003.
- [Result] Boussiotis VA. Molecular and Biochemical Aspects of the PD-1 Checkpoint Pathway. N Engl J Med. 2016 Nov 3;375(18):1767-1778. doi: 10.1056/NEJMra1514296. No abstract available. PMID 27806234
- [Result] Ma W, Gilligan BM, Yuan J, Li T. Current status and perspectives in translational biomarker research for PD-1/PD-L1 immune checkpoint blockade therapy. J Hematol Oncol. 2016 May 27;9(1):47. doi: 10.1186/s13045-016-0277-y. PMID 27234522
- [Result] Havel JJ, Chowell D, Chan TA. The evolving landscape of biomarkers for checkpoint inhibitor immunotherapy. Nat Rev Cancer. 2019 Mar;19(3):133-150. doi: 10.1038/s41568-019-0116-x. PMID 30755690
- [Result] Kitano Y, Yamashita YI, Nakao Y, Itoyama R, Yusa T, Umezaki N, Tsukamoto M, Yamao T, Miyata T, Nakagawa S, Okabe H, Imai K, Chikamoto A, Ishiko T, Baba H. Clinical Significance of PD-L1 Expression in Both Cancer and Stroma Cells of Cholangiocarcinoma Patients. Ann Surg Oncol. 2020 Feb;27(2):599-607. doi: 10.1245/s10434-019-07701-4. Epub 2019 Aug 12. PMID 31407173
- [Result] Neyaz A, Husain N, Kumari S, Gupta S, Shukla S, Arshad S, Anand N, Chaturvedi A. Clinical relevance of PD-L1 expression in gallbladder cancer: a potential target for therapy. Histopathology. 2018 Oct;73(4):622-633. doi: 10.1111/his.13669. Epub 2018 Jul 13. PMID 29882997
- [Result] Ahn S, Lee Y, Kim JW, Lee JC, Hwang JH, Yoon YS, Cho JY, Han HS, Choi Y, Kim H. Programmed cell death ligand-1 (PD-L1) expression in extrahepatic biliary tract cancers: a comparative study using 22C3, SP263 and E1L3N anti-PD-L1 antibodies. Histopathology. 2019 Oct;75(4):526-536. doi: 10.1111/his.13901. Epub 2019 Aug 2. PMID 31081949
- [Result] Kriegsmann M, Roessler S, Kriegsmann K, Renner M, Longuespee R, Albrecht T, Loeffler M, Singer S, Mehrabi A, Vogel MN, Pathil A, Kohler B, Springfeld C, Rupp C, Weiss KH, Goeppert B. Programmed cell death ligand 1 (PD-L1, CD274) in cholangiocarcinoma - correlation with clinicopathological data and comparison of antibodies. BMC Cancer. 2019 Jan 15;19(1):72. doi: 10.1186/s12885-018-5254-0. PMID 30646854
- [Result] Kang J, Yoo C, Jeong JH et al. Efficacy and safety of pembrolizumab in patients with PD-L1 positive advanced biliary tract cancer (BTC): A prospective cohort study. Journal of Clinical Oncology 2019; 37: 4082-4082.
- [Result] Kim RD, Kim DW, Alese OB et al. A phase II study of nivolumab in patients with advanced refractory biliary tract cancers (BTC). Journal of Clinical Oncology 2019; 37: 4097-4097.
- [Result] Smyth MJ, Ngiow SF, Ribas A, Teng MW. Combination cancer immunotherapies tailored to the tumour microenvironment. Nat Rev Clin Oncol. 2016 Mar;13(3):143-58. doi: 10.1038/nrclinonc.2015.209. Epub 2015 Nov 24. PMID 26598942
- [Result] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Result] Ueno M, Ikeda M, Sasaki T, Nagashima F, Mizuno N, Shimizu S, Ikezawa H, Hayata N, Nakajima R, Morizane C. Phase 2 study of lenvatinib monotherapy as second-line treatment in unresectable biliary tract cancer: primary analysis results. BMC Cancer. 2020 Nov 16;20(1):1105. doi: 10.1186/s12885-020-07365-4. PMID 33198671
- [Result] Gunda V, Gigliotti B, Ashry T, Ndishabandi D, McCarthy M, Zhou Z, Amin S, Lee KE, Stork T, Wirth L, Freeman GJ, Alessandrini A, Parangi S. Anti-PD-1/PD-L1 therapy augments lenvatinib's efficacy by favorably altering the immune microenvironment of murine anaplastic thyroid cancer. Int J Cancer. 2019 May 1;144(9):2266-2278. doi: 10.1002/ijc.32041. Epub 2019 Jan 24. PMID 30515783
- [Result] Kato Y, Tabata K, Kimura T, Yachie-Kinoshita A, Ozawa Y, Yamada K, Ito J, Tachino S, Hori Y, Matsuki M, Matsuoka Y, Ghosh S, Kitano H, Nomoto K, Matsui J, Funahashi Y. Lenvatinib plus anti-PD-1 antibody combination treatment activates CD8+ T cells through reduction of tumor-associated macrophage and activation of the interferon pathway. PLoS One. 2019 Feb 27;14(2):e0212513. doi: 10.1371/journal.pone.0212513. eCollection 2019. PMID 30811474
- [Result] Llovet J, Shepard KV, Finn RS et al. 747PA phase Ib trial of lenvatinib (LEN) plus pembrolizumab (PEMBRO) in unresectable hepatocellular carcinoma (uHCC): Updated results. Annals of Oncology 2019; 30.
- [Result] Lin J, Shi W, Zhao S et al. Lenvatinib plus checkpoint inhibitors in patients (pts) with advanced intrahepatic cholangiocarcinoma (ICC): Preliminary data and correlation with next-generation sequencing. Journal of Clinical Oncology 2018; 36: 500-500.
- [Result] Lin J, Yang X, Zhao S et al. 1272PLenvatinib plus PD-1 blockade in advanced bile tract carcinoma. Annals of Oncology 2019; 30.
- [Result] Tang B, Yan X, Sheng X, Si L, Cui C, Kong Y, Mao L, Lian B, Bai X, Wang X, Li S, Zhou L, Yu J, Dai J, Wang K, Hu J, Dong L, Song H, Wu H, Feng H, Yao S, Chi Z, Guo J. Safety and clinical activity with an anti-PD-1 antibody JS001 in advanced melanoma or urologic cancer patients. J Hematol Oncol. 2019 Jan 14;12(1):7. doi: 10.1186/s13045-018-0693-2. PMID 30642373
- [Result] Sheng X, Yan X, Chi Z, Si L, Cui C, Tang B, Li S, Mao L, Lian B, Wang X, Bai X, Zhou L, Kong Y, Dai J, Wang K, Tang X, Zhou H, Wu H, Feng H, Yao S, Flaherty KT, Guo J. Axitinib in Combination With Toripalimab, a Humanized Immunoglobulin G4 Monoclonal Antibody Against Programmed Cell Death-1, in Patients With Metastatic Mucosal Melanoma: An Open-Label Phase IB Trial. J Clin Oncol. 2019 Nov 10;37(32):2987-2999. doi: 10.1200/JCO.19.00210. Epub 2019 Aug 12. PMID 31403867
- [Result] Hodi FS, Ballinger M, Lyons B, Soria JC, Nishino M, Tabernero J, Powles T, Smith D, Hoos A, McKenna C, Beyer U, Rhee I, Fine G, Winslow N, Chen DS, Wolchok JD. Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST): Refining Guidelines to Assess the Clinical Benefit of Cancer Immunotherapy. J Clin Oncol. 2018 Mar 20;36(9):850-858. doi: 10.1200/JCO.2017.75.1644. Epub 2018 Jan 17. PMID 29341833